CLINICAL TRIAL: NCT07011173
Title: Assistance Delivery and Muscle Coordination
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: The Catholic University of America (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: STUDY00006784; 1R15HD114052 (NIH)
Record Dates: First submitted 2025-05-29; First posted 2025-06-08 (Actual); Last update posted 2025-07-23 (Actual); Status verified 2025-07

CONDITIONS: Stroke
Keywords: Stroke; Muscle coordination; Assistance
MeSH Terms: conditions — Stroke; Helping Behavior

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- End-effector assistance followed by exotendon assistance (Experimental)
  Interventions: Device: Exotendon assistance; Device: End-effector assistance
- Exotendon assistance followed by end-effector assistance (Experimental)
  Interventions: Device: Exotendon assistance; Device: End-effector assistance

INTERVENTIONS:
Device: Exotendon assistance — Assistive devices with distinct assistance dynamics
Device: End-effector assistance — Finger will be moved by the actuators connected to the fingertip

SUMMARY:
The experiment will be conducted with 15 chronic stroke survivors and 15 control subjects. Subjects will perform extension movements of the index finger of their more-impaired (stroke) or nondominant (control) hand under two different assistance types: end-effector assistance and exotendon assistance. For each assistance type, unassisted movements will be performed before and after the assistance. Subjects will be randomly assigned into two groups (A and B), who will receive the assistance in a different order. The finger movements and muscle activation patterns will be recorded during movements.

DETAILED DESCRIPTION:
1. Pre-experimental session:

   First, reflective markers will be placed on the dorsum of the hand, i.e., metacarpophalangeal (MCP) and distal/proximal interphalangeal (DIP/PIP) joints of the index finger, index fingertip, MCP of the little finger, and carpometacarpal joint of the middle finger, which will be used to establish a local coordinate system. ten-camera motion capture system (Optitrak Prime X13; NaturalPoint Inc., OR, USA) will be used to record the finger movements.

   Bipolar surface electrodes (Myosystem 14; Noraxon Inc., Scottsdale, AZ) will be placed to record the activity of the following muscles: extensor digitorum communis (EDC), flexor digitorum superficialis (FDS), first dorsal interosseous (FDI), first palmar interosseous (FPI), extensor carpi radialis (ECR), and flexor carpi radialis (FCR) muscles.

   Once the reflective markers and the electromyography (EMG) electrodes are attached, subjects will place their hand in the device. Their forearm will be secured once a comfortable wrist posture for each subject is determined. The location of the pulleys and linear guides will be adjusted to accommodate the forearm posture, determined by the subject-specific wrist angle. Once the fingertip is secured to the end-effector actuator, whose location will then be fixed/locked, they will perform maximum contraction (3-second) of the following muscles, extensor digitorum communis (EDC), flexor digitorum superficialis (FDS), first dorsal interosseous (FDI), extensor carpi radialis (ECR), and flexor carpi radialis (FCR) by performing finger extension, finger flexion, finger abduction, wrist extension, and wrist flexion, during which maximum EMG signals for the target muscles will be obtained. Rest periods of minimum 30-second (or as needed) will be administered between contractions. The fingertip will then be disconnected from the end-effector.
2. Experimental session (1,2):

After rest, subjects will perform finger extension movements with and without assistance. In each session, finger extension task will be performed without assistance in the block 1 (10 trials), followed by the assisted finger extension in the block 2 (15 trials). In the block 3, unassisted finger extension will be performed to gauge residual impact of the motor adaptation by assistance (Fig. 1B).

For group A, session 1 (end-effector assistance) will first be tested, followed by session 2 (exotendon assistance); for group B, the session 2 will be first implemented.

1. Unassisted finger extension: Subjects will extend their index finger from the initial posture (approximately MCP: 45°; PIP: 60°; DIP: 45°) to the fully-extended posture (all angles = 0°).
2. Assisted finger extension (end-effector): The two linear motors will be coordinated to produce a smooth fingertip trajectory for the finger extension. A custom MATLAB program will generate the time-varying movement profiles of the two linear motors that produce the desired fingertip trajectory for each subject in 3 seconds, which are computed from each subject's segment lengths and initial/final postures of the finger extension movement (forward kinematics).
3. Assisted finger extension (exotendon): The two exotendons (extrinsic extensor and intrinsic cables; Fig. 2) will be pulled to assist finger extension movement. Actuation speed of the two linear motors, pulling the extrinsic extensor exotendon (mimicking EDC action) and the intrinsic exotendon (mimicking FDI/FPI action), will be determined from the total excursion of the two exotendons during extension movement, which depends on the subject's finger thickness (i.e., moment arms of the exotendons). The motor speed will be adjusted so that the finger extension movement can be completed in 3 seconds.

In all conditions, a graphical user interface (MATLAB toolbox) will display a timing bar that indicates the timing of the movement initiation and completion (duration: 3 seconds).

ELIGIBILITY:
Inclusion Criteria for stroke survivors:

* Age: 18 - 70 years old
* First-ever unilateral cortical stroke with resultant hemiparesis at least 6 months prior to the experimental testing
* Fugl-Meyer Upper Extremity Section 31 - 55

Exclusion Criteria for both stroke and control:

* Presence of concurrent severe medical illness
* Pain in hand or arm with movements
* Loss of voluntary control of fingers and thumb
* Inability to provide informed consent
* Musculoskeletal injuries (e.g., fracture) or medical complications (e.g., severe cardiovascular disease).

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-11-21 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Muscle activation pattern | Periprocedural
  Coordination of different hand muscles

CONTACTS AND LOCATIONS:
Locations (1):
- Catholic University of America, Washington D.C., District of Columbia, United States

IPD SHARING:
Plan to Share IPD: Undecided
The investigators have not decided how and which part of the data will be shared.